CLINICAL TRIAL: NCT06075095
Title: A Randomised, Placebo-Controlled, Double-Blind, Multi-Centre, 4-week, 3-way Crossover Pharmacodynamic Study to Assess the Equivalence of Budesonide, Glycopyrronium, and Formoterol Fumarate (BGF) Delivered by MDI HFO Compared With BGF Delivered by MDI HFA in Participants With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Investigate the Effect on Lung Function of an Approved COPD Treatment (BGF, With HFA Propellant) Compared to BGF Formulated With a Next-Generation Propellant in Participants 40 to 80 Years of Age With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5985C00002; 2023-506565-57-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Glycopyrrolate; Formoterol Fumarate; 1,3,3,3-tetrafluoropropene

STUDY DESIGN:
Intervention Model Description: This is a phase III, randomised, placebo-controlled, double-blind, multi-centre, 4-week, 3-way crossover pharmacodynamic study to assess the equivalence of BGF MDI HFO compared with BGF MDI HFA in participants with COPD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence 1 (Experimental): Each participant will participate in 3 treatment periods of approximately 4 weeks each (one period for each of 3 study interventions) in the following sequence.
  Sequence 1:
  BGF MDI HFO 320/14.4/9.6 μg BGF MDI HFA 320/14.4/9.6 μg Placebo MDI HFA
  Interventions: Drug: BGF MDI HFO 320/14.4/9.6μg; Drug: BGF MDI HFA 320/14.4/9.6 μg; Drug: Placebo MDI HFA
- Treatment Sequence 2 (Experimental): Each participant will participate in 3 treatment periods of approximately 4 weeks each (one period for each of 3 study interventions) in the following sequence.
  Sequence 2:
  BGF MDI HFO 320/14.4/9.6 μg Placebo MDI HFA BGF MDI HFA 320/14.4/9.6 μg
  Interventions: Drug: BGF MDI HFO 320/14.4/9.6μg; Drug: BGF MDI HFA 320/14.4/9.6 μg; Drug: Placebo MDI HFA
- Treatment Sequence 3 (Experimental): Each participant will participate in 3 treatment periods of approximately 4 weeks each (one period for each of 3 study interventions) in the following sequence.
  Sequence 3:
  BGF MDI HFA 320/14.4/9.6 μg BGF MDI HFO 320/14.4/9.6 μg Placebo MDI HFA
  Interventions: Drug: BGF MDI HFO 320/14.4/9.6μg; Drug: BGF MDI HFA 320/14.4/9.6 μg; Drug: Placebo MDI HFA
- Treatment Sequence 4 (Experimental): Each participant will participate in 3 treatment periods of approximately 4 weeks each (one period for each of 3 study interventions) in the following sequence.
  Sequence 4:
  BGF MDI HFA 320/14.4/9.6 μg Placebo MDI HFA BGF MDI HFO 320/14.4/9.6 μg
  Interventions: Drug: BGF MDI HFO 320/14.4/9.6μg; Drug: BGF MDI HFA 320/14.4/9.6 μg; Drug: Placebo MDI HFA
- Treatment Sequence 5 (Experimental): Each participant will participate in 3 treatment periods of approximately 4 weeks each (one period for each of 3 study interventions) in the following sequence.
  Sequence 5:
  Placebo MDI HFA BGF MDI HFO 320/14.4/9.6 μg BGF MDI HFA 320/14.4/9.6 μg
  Interventions: Drug: BGF MDI HFO 320/14.4/9.6μg; Drug: BGF MDI HFA 320/14.4/9.6 μg; Drug: Placebo MDI HFA
- Treatment Sequence 6 (Experimental): Each participant will participate in 3 treatment periods of approximately 4 weeks each (one period for each of 3 study interventions in the following sequence.
  Sequence 6:
  Placebo MDI HFA BGF MDI HFA 320/14.4/9.6 μg BGF MDI HFO 320/14.4/9.6 μg
  Interventions: Drug: BGF MDI HFO 320/14.4/9.6μg; Drug: BGF MDI HFA 320/14.4/9.6 μg; Drug: Placebo MDI HFA

INTERVENTIONS:
Drug: BGF MDI HFO 320/14.4/9.6μg — Study interventions will be administered orally via MDI as 2 inhalations BID (every morning and evening, approximately 12 hours apart)
  Other Names: Budesonide, Glycopyrronium, and Formoterol Fumarate (BGF); Delivered by MDI HFO (HFO-1234ze)
Drug: BGF MDI HFA 320/14.4/9.6 μg — Study interventions will be administered orally via MDI as 2 inhalations BID (every morning and evening, approximately 12 hours apart):
  Other Names: Budesonide, Glycopyrronium, and Formoterol Fumarate (BGF); Delivered by MDI HFA
Drug: Placebo MDI HFA — Study interventions will be administered orally via MDI as 2 inhalations BID (every morning and evening, approximately 12 hours apart)
  Other Names: Placebo

SUMMARY:
The purpose of this study is to demonstrate that the lung function effect from orally inhaled BGF delivered via HFO propellant is equivalent to the lung function effect from orally inhaled BGF delivered via HFA propellant in participants with COPD. The study duration for each participant will be approximately 15 to 16 weeks and consist of:

1. A screening and placebo run-in period of approximately 2 weeks prior to first dosing
2. Three treatment periods of approximately 4 weeks each (one period for each of 3 study interventions)
3. A final safety follow-up visit via telephone contact approximately 1 to 2 weeks after the final dose administration Participants will be provided with rescue SABA (albuterol or salbutamol) to be used as needed throughout the study. Participants will attend in-clinic study visits approximately weekly during the screening/run-in period (Visits 1, 2, and 3), then every 4 weeks (Visits 4, 5, and 6) to receive take-home study treatment, measure their lung function, and assess their health and safety

DETAILED DESCRIPTION:
This is a phase III, randomised, placebo-controlled, double-blind, multi-centre, 4-week, 3-way crossover pharmacodynamic study to assess the equivalence of BGF MDI HFO compared with BGF MDI HFA in participants with COPD. To demonstrate assay sensitivity, BGF MDI HFA will be compared to placebo MDI HFA for superiority in lung function, both pre- and post-dose.

Eligible participants are between 40 and 80 years of age, inclusive, who have an established clinical history of COPD as defined by the ATS/ERS. Participants are required to have an FEV1/FVC ratio of < 0.70, have a post-bronchodilator FEV1 ≥ 40% and < 80% predicted normal value, have a blood eosinophil count < 300 cells/μL, and be current or former cigarette smokers with a history of at least 10 pack-years. Participants must not have had a COPD exacerbation treated with oral corticosteroids or antibiotics within 4 months prior to initiation of screening, and must not have had a COPD exacerbation that required hospitalisation within 12 months prior to initiation of screening. Eligible participants are those on treatment with LABA, LAMA, LAMA/LABA (open or fixed-dose combination), ICS/LABA (open or fixed-dose combination) inhaled maintenance therapies, or SABA, SAMA, or SAMA/SABA scheduled or as-needed inhaled therapies, or who are naïve to COPD therapy.

This study will be conducted at approximately 95 sites globally. After screening, participants will be randomised 1:1:1:1:1:1 to receive study interventions in one of 6 possible treatment sequences.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Age

1. Participants must be 40 to 80 years inclusive at the time of signing the ICF. Type of Participant and Disease Characteristics
2. Participants who have a documented history of physician-diagnosed COPD as defined by the ATS/ERS (Celli et al 2004).
3. Participants who have been receiving LABA, LAMA, LAMA/LABA, or ICS/LABA inhaled maintenance therapies for the management of their COPD for at least 4 weeks prior to Visit 1, OR Participants who have been receiving SABA, SAMA, or SABA/SAMA either scheduled or as needed for at least 4 weeks prior to Visit 1, OR Participants who are COPD treatment-naïve or have not received previously prescribed COPD treatment in the 4 weeks prior to Visit 1.
4. At Visit 1: Participants with a blood eosinophil count < 300 cells/μL.
5. At Visit 1: Participants with a pre-bronchodilator FEV1 of < 80% predicted normal.
6. At Visit 2: Participants with a post-bronchodilator FEV1/FVC ratio of < 0.70 and a postbronchodilator FEV1 of ≥ 40% to < 80% predicted normal.
7. At Visit 3 (TP 1 Day 1): Participants with a pre-dose FEV1 of < 80% predicted normal that is within ± 20% or 200 mL of their Visit 2 pre-bronchodilator FEV1 and an FEV1/FVC ratio of < 0.70.
8. Current or former smokers with a history of at least 10 pack-years of tobacco smoking

<!-- -->

1. pack-year = 20 cigarettes smoked per day for one year). 9 Participants who are willing and, in the opinion of the Investigator, able to adjust current COPD therapy, as required by the protocol. Sex and Contraceptive/Barrier Requirements 10 Females must not be of childbearing potential or must use a form of highly effective birth control as defined below:

   * Females not of childbearing potential are defined as females who are either permanently sterilised (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or postmenopausal. Females will be considered postmenopausal if they have been amenorrhoeic for 52 weeks (12 months) prior to the planned date of randomisation without an alternative medical cause. The following age-specific requirements apply:

     * Females < 50 years old would be considered postmenopausal if they have been amenorrhoeic for 52 weeks (12 months) or more following cessation of exogenous hormonal treatment with FSH levels in the postmenopausal range.
     * Females ≥ 50 years old would be considered postmenopausal if they have been amenorrhoeic for 52 weeks (12 months) or more following cessation of all exogenous hormonal treatment.
   * Female participants of childbearing potential must use one highly effective form of birth control. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly.

   All FOCBP who are sexually active with a non-sterilised male partner must agree to use one highly effective method of birth control, as defined below, from enrolment throughout the study and until at least 14 days after the last dose of study intervention. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational [15:32] Łubian, Dominika amenorrhoea method are not acceptable methods of contraception. Female condom and male condom should not be used together.

   - All FOCBP must have a negative serum pregnancy test result at Visit 1.

   - Females < 50 years of age with amenorrhoea for at least 12 months without an alternative medical cause must have a serum FSH test at Visit 1.
   * Highly effective birth control methods are listed below:

     - Total sexual abstinence is an acceptable method provided it is the preferred and usual lifestyle of the participant (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study interventions).

     - Combined (oestrogen and progestogen-containing) hormonal contraception associated with inhibition of ovulation:

     o Oral

     o Intravaginal

     o Transdermal
     * Progestogen-only hormonal contraception associated with inhibition of ovulation: o Oral

       o Injectable
       * Implantable
     * Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
     * Bilateral tubal occlusion
     * Male partner sterilisation/vasectomy with documentation of azoospermia prior to the female participant's entry into the study, and this male is the sole partner for that participant. The documentation on male sterility can come from the site personnel's review of participant's medical records, medical examination and/or semen analysis or medical history interview provided by her or her partner. Informed Consent 11 Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

   Other Inclusion Criteria 12 Participants with calculated eGFR > 30 mL/min/1.73 m2 using the CKD-EPI formula.

13 Participants who demonstrate acceptable MDI administration and spirometry techniques.

14 Participants who remain compliant with placebo run-in administrations, defined as ≥ 80% of planned doses over the last 7 days prior to Visit 3, based on ePRO diary data.

15 Participants who are willing to remain at the study centre as required per protocol to complete all visit assessments.

Exclusion Criteria:

Medical Conditions

1. Confirmed diagnosis of asthma, in the opinion of the Investigator based on thorough review of medical history and medical records.
2. COPD due to α1-antitrypsin deficiency.
3. A COPD exacerbation treated with systemic corticosteroids or antibiotics within 4 months prior to Visit 1 or during the Screening Period.
4. A COPD exacerbation that required hospitalisation within 12 months prior to Visit 1 or during the Screening Period.
5. A respiratory infection ending within 4 weeks prior to Visit 1 or beginning or ending during the Screening Period, per the Investigator's judgement.
6. Life-threatening COPD (eg, need for mechanical ventilation) at any time prior to Visit 1 or during the Screening Period.
7. A SARS-CoV-2 infection in the 8 weeks prior to Visit 1 or during the Screening Period, or that required hospitalisation at any time prior to Visit 1 or during the Screening Period.
8. Sleep apnoea that, in the opinion of the Investigator, is uncontrolled.
9. Other respiratory disorders including, but not limited to, known active tuberculosis, lung cancer, cystic fibrosis, significant bronchiectasis (high-resolution CT evidence of bronchiectasis that causes repeated acute exacerbations), severe neurological disorders affecting control of the upper airway, sarcoidosis, primary ciliary dyskinesia, idiopathic interstitial pulmonary fibrosis, primary pulmonary hypertension, or pulmonary thromboembolic disease.
10. Significant or unstable ischaemic heart disease, arrhythmia, cardiomyopathy, heart failure, uncontrolled hypertension as defined by the Investigator, or any other relevant cardiovascular disorder as judged by the Investigator.
11. Diagnosis of narrow-angle glaucoma that has not been adequately treated, or a change in vision that may be relevant, in the opinion of the Investigator.

    Note: All medications approved for control of intraocular pressures are allowed, including topical ophthalmic nonselective beta-blockers and prostaglandin analogues.
12. Symptomatic prostatic hypertrophy or bladder neck obstruction/urinary retention that, in the opinion of the Investigator, is clinically significant.
13. Unresectable cancer that has not been in complete remission for at least 5 years prior to Visit 1. Note: Squamous cell and basal cell carcinomas of the skin are allowed.
14. Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular, hepatic, renal, haematological, neurological, endocrine, gastrointestinal, or pulmonary. Immune deficiency disorders (ie, HIV infection) should be excluded even if controlled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the participant at risk through participation, or that could affect the efficacy or safety analysis if the disease/condition is exacerbated during the study.
15. Participants with a known hypersensitivity to beta2-agonists, muscarinic antagonists, or corticosteroids, or any component of the MDI.
16. Known history of drug or alcohol abuse within 12 months of Visit 1 or known abuse at any time during the study.
17. History of QT prolongation associated with another medication that required discontinuation of that medication.

    Prior/Concomitant Therapy
18. Unable to abstain from short-acting bronchodilators within 6 hours prior to lung function testing at each study visit.
19. Pulmonary resection or lung volume reduction surgery during the 6 months prior to Visit 1 (ie, lobectomy, bronchoscopic lung volume reduction [endobronchial blockers, airway bypass, endobronchial valves, thermal vapour ablation, biological sealants, and airway implants]).
20. Long-term-oxygen therapy or nocturnal oxygen therapy required for greater than 15 hours per day.

    Note: As-needed oxygen use is allowed.
21. Trans-urethral resection of the prostate or full resection of the prostate within 6 months prior to Visit 1.
22. Unable to abstain from any protocol-defined prohibited medications during the Screening or Treatment Periods (see Section 6.9).
23. Use of any herbal products by either inhalation or nebuliser within 2 weeks prior to Visit 1 or refusal to stop use for the duration of the study.

    Prior/Concurrent Clinical Study Experience
24. Participation in another clinical study with a study intervention administered within 30 days or 5 half-lives, whichever is longer, prior to Visit 1.

    Diagnostic Assessments
25. Participants with ECG QTcF interval > 480 milliseconds.
26. Participants with high-degree atrioventricular block II or III, or with sinus node dysfunction with clinically significant pauses who are not treated with pacemaker.
27. Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs, or ECG which, in the opinion of the Investigator, may put the participant at risk because of their participation in the study.

    Other Exclusions
28. Planned hospitalisation during the study.
29. Involvement in the planning or conduct of the study (applies to both AstraZeneca staff and staff at the study sites).
30. Study Investigators, sub-Investigators, coordinators, and their employees or immediate family members.
31. Judgement by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
32. Previous randomisation in the present study.
33. For women only: currently pregnant (confirmed with positive pregnancy test), breastfeeding, or planned pregnancy during the study, or FOCBP not using acceptable contraception measures.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Changes in FEV1 AUC (0-4) | Change from baseline at Day 29
  To assess the equivalence of BGF MDI HFO relative to BGF MDI HFA on lung function in participants with COPD
Change in morning pre-dose trough FEV1 | Change from baseline at Day 29
  To assess the equivalence of BGF MDI HFO relative to BGF MDI HFA on lung function in participants with COPD
Changes in FEV1 AUC (0-4) | Change from baseline at Day 29
  To demonstrate assay sensitivity via superiority of BGF MDI HFA relative to placebo MDI HFA on lung function in participants with COPD
Change in morning pre-dose trough FEV1 | Change from baseline at Day 29
  To demonstrate assay sensitivity via superiority of BGF MDI HFA relative to placebo MDI HFA on lung function in participants with COPD

OTHER OUTCOMES:
Number (and percentage) of participants with adverse Events | Over 16 weeks and per treatment group per 4 weeks treatment period
  To assess the safety and tolerability of BGF MDI HFO compared to BGF MDI HFA in participants with COPD
Number (and percentage) of participants with with potentially clinically significant changes in Blood Pressure | Over 16 weeks and per treatment group per 4 weeks treatment period
  To assess the safety and tolerability of BGF MDI HFO compared to BGF MDI HFA in participants with COPD
Number (and percentage) of participants with potentially clinically significant changes in pulse rate | Over 16 weeks and per treatment group per 4 weeks treatment period
  To assess the safety and tolerability of BGF MDI HFO compared to BGF MDI HFA in participants with COPD
Changes in FEV1 AUC (0-4) | Change from baseline at TP 1 Day 1
  To determine responsiveness to study intervention for TP 1
Time to onset of action | Change from baseline at TP 1 Day 1
  Time to onset defined as the first post-dose timepoint where the mean change from baseline in FEV1 exceeds 100 mL on TP 1 Day 1
Changes in FEV1 AUC (0-4) | Change from baseline at Day 29
  To assess superiority of BGF MDI HFO relative to placebo MDI HFA on lung function, pre- and post-dose, in participants with COPD
Change in morning pre-dose trough FEV1 | Change from baseline at Day 29
  To assess superiority of BGF MDI HFO relative to placebo MDI HFA on lung function, pre- and post-dose, in participants with COPD

CONTACTS AND LOCATIONS:
Locations (82):
- United States (19):
  - Research Site, Sheffield, Alabama
  - Research Site, Clearwater, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Rincon, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, The Bronx, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Dublin, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Gaffney, South Carolina
  - Research Site, Boerne, Texas
  - Research Site, El Paso, Texas
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, San Fernando
- Bulgaria (8):
  - Research Site, Burgas
  - Research Site, Pernik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Vratsa
- Canada (5):
  - Research Site, Truro, Nova Scotia
  - Research Site, Burlington, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
- Hungary (5):
  - Research Site, Balassagyarmat
  - Research Site, Hajdúnánás
  - Research Site, Mosonmagyaróvár
  - Research Site, Pécs
  - Research Site, Püspökladány
- India (6):
  - Research Site, Ajmer
  - Research Site, Aligarh
  - Research Site, Coimbatore
  - Research Site, Jaipur
  - Research Site, Kanpur
  - Research Site, Surat
- Malaysia (4):
  - Research Site, George Town
  - Research Site, Ipoh
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Terengganu
- Mexico (5):
  - Research Site, Benito Juárez
  - Research Site, Chihuahua City
  - Research Site, Cuernavaca
  - Research Site, Monterrey
  - Research Site, Zapopan
- Philippines (3):
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Quezon City
- Poland (3):
  - Research Site, Bialystok
  - Research Site, Chęciny
  - Research Site, Lublin
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Ulsan
- Thailand (4):
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Dinar
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kayseri
- Vietnam (7):
  - Research Site, Can Tho
  - Research Site, Da Nang
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home